CLINICAL TRIAL: NCT01277380
Title: Analysis of the Results From Influenza Rapid Test A Positive and H1N1 Real Time RT-PCR
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Taipei Medical University WanFang Hospital (Other)
Responsible Party: Giueng-Chueng Wang, Laboratory Medicine, Wanfang Hospital
Other Study IDs: 99029
Record Dates: First submitted 2011-01-12; First posted 2011-01-14 (Estimated); Last update posted 2011-01-14 (Estimated); Status verified 2011-01

CONDITIONS: H1N1 Influenza Virus
Keywords: H1N1 Influenza virus; swine flu; Real Time RT-PCR
MeSH Terms: conditions — Orthomyxoviridae Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Experimental Group
- Control Group
- Negative control group

SUMMARY:
The first outbreak of a new H1N1 influenza pandemic originated in the North America in April 2009. As of July 1, 2009, a total of 77,201 cases were accumulated in 103 countries around the world and the mortality rate of was about 0.43%. Alignment and analysis on gene sequences of the new H1N1 influenza virus found that it contains extremely homologous gene composition with that of the swine influenza viruses (swine flu) identified in Europe and North America in last century. Thus the virus strain was later renamed as a novel influenza H1N1. In general, the symptoms caused by the new influenza H1N1 infection was very similar to those resulted from seasonal influenza viral infection. Thus, it is difficult to distinguish the various influenza strains responsible for the infections only by clinical appearance. To compare the accuracy, specificity and sensitivity and speed in identifying the new influenza H1N1 in suspected cases, the investigators extracted RNA from influenza A-positive reactive specimens identified by a Influenza Rapid Test, for a Real-time PCR method to further detect the presence of swine H1 gene. In addition, the titer of H1N1 virus, the color development on the test stripe and clinical symptoms in patients were significantly associated. Finally, Real-time PCR products were subjected to sequence determination to explore potential new influenza pathogenicity, transmissibility and drug usage.

ELIGIBILITY:
Inclusion Criteria:

* Influenza Rapid Test Influenza A(+) B(-)
* Influenza Rapid Test Influenza A(+) B(+)
* Influenza Rapid Test Influenza A(-) B(-) was negative control

Exclusion Criteria:

* Influenza Rapid Test Influenza A(-) B(+)

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: H1N1 Influenza
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2010-08; Study Completion 2011-08 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Giueng-Chueng Wang, Principal Investigator — Taipei Medical University WanFang Hospital
Locations (1):
- Taipei Medical University - WanFang Hospital, Taipei, Taiwan